CLINICAL TRIAL: NCT06642168
Title: Registre Prospectif Français Des Morts Subites Chez Des Sportifs Jeunes
Brief Title: Sudden Cardiac Arrest Related to Sport in Young and Value of the Genetic Assessment: a French Prospective Register
Acronym: RESOUDRE
Status: Recruiting | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC19_8911_RESOUDRE
Record Dates: First submitted 2024-10-08; First posted 2024-10-15 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Sudden Cardiac Arrest; Sudden Cardiac Death
Keywords: Sport related sudden cardiac arrest; Sport related sudden cardiac death; Young athlete; Etiological Diagnosis; Autopsy; Genetic; Toxicology; Hereditary Cardiac disease; Prevention
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Victims of sport-related sudden cardiac arrest (SCA) : resuscitated SCA and non-resuscitated SCA: Following a sport-related sudden cardiac arrest (SCA), resuscitation attempts are frequently made due to the high likelihood of witnesses at the scene. These resuscitation efforts are successful in more than 40% of cases. The study population will therefore be divided into two groups: a group of resuscitated SCA victims (SCA group) and a group of non-resuscitated or unsuccessfully resuscitated victims (SCD group).
  The RESOUDRE study is an observational study focusing on individuals who have experienced SCA. Depending on the outcome-whether the individual survives or not-the etiological assessment will differ. While the study design refers to two distinct groups for clarity, they represent a single population, and no statistical comparison between the two groups will be made.
  Interventions: Genetic: Whole exome sequencing to detect myocardial genetic mutations (SCA group only)

INTERVENTIONS:
Genetic: Whole exome sequencing to detect myocardial genetic mutations (SCA group only) — Whole exome sequencing to detect myocardial genetic mutations

SUMMARY:
The increased risk of sudden cardiac arrest (SCA) or sudden cardiac death (SCD) related to vigorous physical activity is well-documented. Currently, for young victims (under 35 years) of SCA/SCD, no etiology is found in 40 to 50% of cases after a standard medical assessment, leading to two important consequences. For the victim's family, it is difficult to understand and accept this tragic event, and the risk of it occurring in another family member is a source of concern. Medically, the absence of a known cause limits the ability to effectively prevent such events.

The RESOUDRE study will be a national, prospective, observational registry of young victims (12-35 years) of sports-related SCA/SCD. All cases will undergo the recommended etiological assessment, including autopsy for SCA cases, along with whole exome genetic analysis and toxicological testing. In the event a genetic pathology is identified, a genetic evaluation will be offered to other family members, and appropriate medical care will be provided if necessary. The results of this study could significantly reduce the number of unexplained sport-related SCA/SCD cases and aid in preventing these incidents among affected families.

DETAILED DESCRIPTION:
Background:

The beneficial effects of moderate physical activity on health are well-established. However, it is also well-proven that intense sports participation increases the risk of cardiovascular events by 2.4 to 4.5 times before the age of 35 in individuals with known or unknown heart conditions. Sudden cardiac arrest (SCA), sometimes leading to sudden cardiac death (SCD), is the most dramatic event linked to sports.

Before the age of 35, sports-related SCA/SCD is rare, occurring in 0.7 to 2.7 per 100,000 athletes, which amounts to approximately 80 cases per year according to two French prospective studies. Despite its rarity, these events are often traumatic and highly publicized, presenting a significant public health and safety concern. Non-traumatic sports-related SCA/SCD is primarily of cardiovascular origin, irrespective of the level of sports participation. In most cases, SCA results from ventricular arrhythmia caused by known or undiagnosed arrhythmogenic cardiovascular disease, which varies by the victim's age. After the age of 35, atheromatous coronary artery disease accounts for 80-85% of cases. However, before the age of 35, a wider range of etiologies are observed. Arrhythmogenic genetic heart diseases-structural (e.g., arrhythmogenic right ventricular cardiomyopathy and hypertrophic cardiomyopathy) or non-structural (e.g., channelopathies)-are the most frequent causes. Congenital abnormalities, particularly anomalous connection of coronary artery, represent the second most common cause. Acquired heart diseases, such as fibrous scars (mainly post-myocarditis) and atheromatous coronary lesions, are less frequently involved. In this younger population, classical autopsy often fails to determine the cause in more than 40% of cases, leading to the term "sudden arrhythmic syndrome".

Few prospective studies have combined classical autopsy with systematic genetic analysis to identify the cause of SCA/SCD in the general young population, with no specific link to sports. One Australian study demonstrated the value of genetic testing, identifying a "clinically relevant" cardiac genetic variant for sudden death in 27% of cases. Moreover, the same pathology was identified in 13% of relatives of the victims who underwent clinical and genetic screening. Another small Swedish study (n=15), focusing specifically on channelopathies in cases of negative autopsies, revealed the disease in 40% of victims' families through genetic analysis.

Additionally, the role of acute or chronic toxic substance intake has been suggested, albeit without formal proof, as a factor promoting sports-related SCA/SCD. Toxicological screening is thus recommended as part of the etiological assessment. Including toxicological analysis alongside other etiological evaluations could help clarify the impact of illicit substances on sports-related SCA/SCD.

Justifications for the Study:

No prospective study has systematically combined the recommended hospital assessment in cases of successful resuscitation or the recommended medical autopsy in the event of death with global genetic and toxicological analyses in victims of sports-related SCA/SCD.

This combined approach is justified for several reasons. First, it would enhance our understanding of the etiologies of these events. Notably, so-called idiopathic left ventricular hypertrophy is found in more than 10% of sports-related SCD cases following classical autopsies. Further genetic exploration could help determine whether these anatomical forms are pathological. Additionally, many arrhythmic cardiac diseases are associated with an elevated risk of sports-related SCA/SCD. While arrhythmogenic right ventricular cardiomyopathy is well-documented, other forms of disease are characterized by areas of fibrosis or fatty infiltration in the myocardium, often due to genetic mutations affecting intercellular desmosomes. Comprehensive genetic testing, including whole exome sequencing, could clarify the contribution of various arrhythmogenic heart diseases to unexplained sports-related SCA/SCD.

Improving this knowledge will benefit ongoing discussions about enhancing the content and effectiveness of pre-participation screening for athletes. Moreover, identifying the cause of SCA/SCD is critical for the victims and their families. Understanding the cause may help families come to terms with the event and assist in preventing recurrence for successfully resuscitated individuals. Furthermore, since most hereditary heart diseases follow an autosomal dominant inheritance pattern, each first-degree relative has a 50% chance of carrying the same genetic mutation. Predictive testing, clinical assessment, and, if necessary, preventive treatment can be offered to these family members to reduce the risk of arrhythmic events.

Statistical Analysis:

Data analyses will be performed using specialized software, with a significance threshold set at 5%. Hypotheses will be formulated bilaterally.

A descriptive analysis of the collected population data will be conducted. Qualitative variables will be presented as numbers and percentages, while quantitative variables will be described using the mean, standard deviation, median, interquartile range, minimum, and maximum values.

For the primary analysis of the main outcome, the cause of sports-related SCA/SCD will be described in terms of numbers and percentages, along with the corresponding 95% confidence intervals.

For the secondary analyses, the judgment criteria, both overall and by vital status (survived or deceased), will be described in numbers and percentages, with 95% confidence intervals.

ELIGIBILITY:
Inclusion Criteria:

* Victims of SCA:

  * Aged between 12 and 35 years
  * No known cardiovascular pathology
  * Experienced a sudden and non-traumatic SCA during or within one hour of participating in sports activities (leisure, training, or competition)
  * For resuscitated victims (SCA group): A person or legal representative who does not oppose participation in the research after being informed about the study (including individuals, organs, or authorities responsible for assisting or representing them if they are unable to express their wishes).
  * For non-resuscitated victims (SCD group): A person who has not formally objected to the reuse of their medical data during their lifetime.
* First-Degree Relatives:

  * A person or legal representative who does not oppose participation in the research after being informed about the study (including individuals, bodies, or authorities responsible for assisting or representing them if they are unable to express their wishes).

Non-Inclusion Criteria:

* For resuscitated SCA cases, individuals weighing less than 20 kg
* Victims or legal representatives who are subject to legal protection or deprived of their liberty

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study will include French victims of sports-related SCA/SCD between the ages of 12 and 35, as well as their first-degree relatives over 12 years of age, when applicable.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-10-11 (Actual); Primary Completion 2028-01-11 (Estimated); Study Completion 2028-01-11 (Estimated)

PRIMARY OUTCOMES:
Identification of the Cause of Sports-Related Cardiorespiratory Arrest in a Young, Healthy Population | Through study completion, approximately 39 months
  The results for each identified cause of sports-related cardiorespiratory arrest will be presented as the total number of cases (n) and the percentage of the total cases. A 95% confidence interval will also be provided.

SECONDARY OUTCOMES:
Evaluation of the Contribution of Medical Autopsy in Identifying the Etiology of Sports-Related SCA | 3 to 6 months after the event
  Results will be presented as the total number of cases (n) and the percentage of the total cases, with a 95% confidence interval.
Evaluation of the Contribution of Classical Genetic Analysis in Identifying the Etiology of Sports-Related Cardiorespiratory Arrest | 3 to 6 months after the event
  The results will be presented as the total number of cases (n) and the percentage of the total cases, with a 95% confidence interval.
Evaluation of the Contribution of Whole Exome Sequencing in Identifying the Etiology of Sports-Related Cardiorespiratory Arrest | 24 to 30 months after the event
  Results will be presented as the total number of cases (n) and the percentage of the total cases, with a 95% confidence interval.
Evaluation of the Contribution of Toxicological Analysis in Identifying the Etiology of Sports-Related Cardiorespiratory Arrest | 3 to 6 months after the event
  Results will be presented as the total number of cases (n) and the percentage of the total cases, with a 95% confidence interval.
Evaluation of the Familial Transmission of Hereditary Cardiovascular Pathologies Detected | 3 to 12 months after the event.
  Results will be presented as the total number of cases (n) and the percentage of the total cases, with a 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric SCHNELL, Principal Investigator — Study Principal Investigator
Locations (26):
- France (26):
  - APHP Hôpital Bichat, Paris, France
  - APHP Hôpital Européen Georges Pompidou, Paris, France
  - CHU Rennes, Rennes, France
  - CHRU Besançon, Besançon
  - CHU Bordeaux, Bordeaux
  - CHU Brest, Brest
  - CHU Caen, Caen
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - APHP Hôpital Henri-Mondor, Créteil
  - CHU Dijon Bourgogne, Dijon
  - CHU de Grenoble Alpes, Grenoble
  - CHRU Lille, Lille
  - Hospices Civils de Lyon, Lyon
  - APHM Hôpitaux universitaires de Marseille, Marseille
  - CHRU Montpellier, Montpellier
  - CHRU Nancy, Nancy
  - CHU Nantes, Nantes
  - CHU de Nice, Nice
  - APHP Hôpital Pitié-Salpêtrière, Paris
  - CHU Poitiers, Poitiers
  - CHU Reims, Reims
  - CHU Rouen, Rouen
  - CHU Saint-Etienne, Saint-Etienne
  - CHRU Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse
  - CHRU Tours, Tours

IPD SHARING:
Plan to Share IPD: Undecided